CLINICAL TRIAL: NCT05809206
Title: Gluteus Maximus Versus Gluteus Medius Strength On Back Muscles Performance In Patients With Sacroiliac Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Abd El moneim Mahmoud Gomma, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Reham_Gomma_PhD
Record Dates: First submitted 2023-03-17; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Sacroiliac Joint Dysfunction
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glutes maximus Strengthening group (Experimental): Twenty patients received Strengthening exercises for Glutes maximus muscle and conventional physical therapy (corrective exercises and ultrasound).
  Interventions: Other: Glutes maximus strength protocol; Other: Corrective Exercises; Device: Ultrasound
- Glutes Medius Strengthening group (Experimental): Twenty patients received Strengthening exercises for Glutes medius muscle and conventional physical therapy (corrective Exercises and therapeutic ultrasound (US).
  Interventions: Other: Gluteus medius strength program; Other: Corrective Exercises; Device: Ultrasound
- Conventional treatment group (Active Comparator): Twenty Patients received conventional therapy (corrective exercises and ultrasound).
  Interventions: Other: Corrective Exercises; Device: Ultrasound

INTERVENTIONS:
Other: Glutes maximus strength protocol — The subjects attended physical therapy two times. Per week for a total of 10 visits. Each session lasted approximately 30 minutes. In the first five sessions, subjects performed the following exercises to strengthen the gluteus maximus: bilateral bridge, unilateral bridge, and non-weight-bearing hip extension in prone with the knee flexed at 90 degrees. In the next five sessions, abduction and external rotation in a quadruped ("fire hydrant" exercise) and weight-bearing hip extension (known as "deadlift" exercise) were added. Each exercise was performed for 10 repetitions. Elastic resistance was added to the fire hydrant, hip extension in prone and dead lift exercises to allow each subject to perform at a 10-repetition maximum. The resistance for each subject was adjusted weekly as needed. The exercise program was performed under direct supervision only during the physical therapy sessions.
  Arms: Glutes maximus Strengthening group
Other: Gluteus medius strength program — Strengthening exercises for Gluteus Medius subdivisions:
  The anterior GMED exercise: side lying abduction exercise The middle GMED exercise: wall press Exercise The posterior GMED exercise: was the pelvic drop exercise
  Arms: Glutes Medius Strengthening group
Other: Corrective Exercises — The following low back corrective exercises were given:
  To stretch the tight lower back muscles: Seated Forward Bend and Full Squat held for 5 sec and Repeated for 3 times, once a day.
  To strengthen the weak lower abdomen: Draw in and Reverse Crunch 3 seconds, repeated 5 times, once a day.
  To stretch the tight hip flexors: held for 10-15 seconds repeated 5 times on both legs, once a day.
  To stretch the tight quadriceps: held for 3 seconds, repeated 5 times on each side, once a day.
  To strengthen weak hamstrings: Kick Butts 2 sec, repeated 8 times, once a day.
Device: Ultrasound — US was administered in continuous mode at PSIS with patient in prone lying position, with a frequency of 1 MHz and intensity of 0.8 W/cm2 for 5 minutes every alternating day

SUMMARY:
This study will be conducted to compare between the effect of glutes maximus and glutes medius muscles strength on back muscle performance in patients with Sacroiliac joint dysfunction.

DETAILED DESCRIPTION:
The purposes of this study are:

1. To investigate the effect of Gluteus maximus strengthening exercises and Gluteus medius strengthening exercises on back pain in patient with Sacroiliac joint dysfunction
2. To investigate the effect of Gluteus maximus strengthening exercises and Gluteus medius strengthening exercises on back muscle performance in patients with Sacroiliac joint dysfunction
3. To investigate the effects of Gluteus maximus strengthening exercises and Gluteus medius strengthening exercises on function in patient with Sacroiliac joint Dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Age from 25-40 years.
* Patients with chronic lumbopelvic pain (more than 12 weeks) and clinical test positive for SIJD.
* The pain distribution and tenderness on palpation under the posterior superior iliac spine (PSIS) are reliable signs that the SIJ is the source of pain.
* Complaint of unilateral pain rather than bilateral pain is also considered more likely to be coming from an SIJ.
* Patients willing and able to participate in an exercise program safely and without cognitive impairments that would limit their participation.

Exclusion Criteria:

* Neurological disorder, psychosomatic disorder
* Tumor.
* Infection condition.
* Recent surgeries.
* Pregnancy.
* Back pain referred from organic cause.
* Osteoporosis and bone disease (induced or idiopathic).

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-10 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in the peak torque of back muscles | at baseline and after 5 weeks of intervention
  By using isokinetic dynamometer, and the unit of of measurement will be (Kg).
Assessing the change in pain threshold | at baseline and after 5 weeks of intervention
  by using Traditional pressure algometers are ideal for measuring pressure pain threshold (PPTs) of superficial muscles and bony landmarks. Pressure pain threshold has been defined as the lowest stimulus intensity at which a subject perceives mechanical pain
Assessing the change in Functional ability level | at baseline and after 5 weeks of intervention
  By using Modified Oswestry Disability Questionnaire (MODQ). The Oswestry Low Back Pain Disability Questionnaire Arabic version will be used to measure disability caused by low back pain in the general population. It consists of 10 questions each consisting of six alternatives. Every question is scored from 0-5 and a percentage are formulated as a result of the sum of the scores.
Assessing the change in pain intensity | at baseline and after 5 weeks of intervention
  By using visual analogue scale (VAS). This scale will be used to measure the intensity of pain. It has been graded as a 10-cm line, which was used for measuring the intensity of perceived pain. In this scale, zero represents the absence of pain, 1-3 shows mild pain, 4-6 denotes moderate pain, and 7-10 indicates severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Reham Abd El-Moneim, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physica therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided